CLINICAL TRIAL: NCT03363776
Title: Phase 1/2a First in Human Study of BMS-986277 Administered Alone and in Combination With Nivolumab in Advanced Epithelial Tumors
Brief Title: An Investigational Immuno-Therapy Study of Experimental Medication BMS-986277 Given Alone and in Combination With Nivolumab in Epithelial Cancers
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Business objectives have changed
Sponsor: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CA034-001; 2017-002199-24 (EudraCT Number)
Record Dates: First submitted 2017-12-01; First posted 2017-12-06 (Actual); Results first posted 2020-12-19 (Actual); Last update posted 2020-12-19 (Actual); Status verified 2020-11

CONDITIONS: Cancer
MeSH Terms: conditions — Neoplasms | interventions — Nivolumab

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Monotherapy (Experimental): BMS-986277 administered alone
  Interventions: Biological: BMS-986277
- Combination Dose Escalation Therapy (Experimental): BMS-986277 administered in combination with Nivolumab
  Interventions: Biological: BMS-986277; Biological: Nivolumab
- Combination Expansion Therapy (Experimental): BMS-986277 monotherapy with option for subsequent Nivolumab therapy
  Interventions: Biological: BMS-986277; Biological: Nivolumab

INTERVENTIONS:
Biological: BMS-986277 — Specified dose on specified days
Biological: Nivolumab — Specified dose on specified days
  Other Names: Opdivo; BMS-963558
  Arms: Combination Dose Escalation Therapy; Combination Expansion Therapy

SUMMARY:
The purpose of this study is to investigate experimental medication BMS-986277 given alone and in combination with Nivolumab in patients with epithelial cancers.

ELIGIBILITY:
For more information regarding Bristol-Myers Squibb Clinical Trial participation, please visit www.BMSStudyConnect.com

Inclusion Criteria:

* Histological or cytological confirmation of metastatic and/or unresectable metastatic colorectal, prostate, pancreatic, breast, ovarian, or urothelial carcinoma with measureable disease for solid tumors per RECIST v1.1 and for prostate carcinoma per PCWG3
* Presence of at least 2 lesions: at least one with measurable disease as defined by RECIST v1.1 for solid tumors and by PCWG3 for prostate carcinoma for response assessment; at least 1 lesion must be accessible for biopsy in addition to the target lesion
* Participants must have received, and then progressed or been intolerant to, at least 1 standard treatment regimen in the advanced or metastatic setting, if such a therapy exists, and have been considered for all other potentially efficacious therapies prior to enrollment
* ECOG performance status less than or equal to 2

Exclusion Criteria:

* Participants with active central nervous system (CNS) metastases, untreated CNS metastases, or with the CNS as the only site of disease
* Participants with carcinomatous meningitis
* Cytotoxic agents, unless at least 4 weeks have elapsed from last dose of prior anti-cancer therapy and initiation of study treatment
* Participants with active, known, or suspected autoimmune disease

Other protocol defined inclusion/exclusion criteria could apply

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2017-12-06 (Actual); Primary Completion 2019-11-22 (Actual); Study Completion 2019-11-22 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (3):
- Sanford Research, Sioux Falls, South Dakota, United States
- Canada (2):
  - Local Institution, Ottawa, Ontario
  - Princess Margaret Cancer Centre, Toronto, Ontario

REFERENCES:
- See also: BMS Clinical Trial Information — https://www.bms.com/researchers-and-partners/clinical-trials-and-research.html
- See also: BMS Clinical Trial Patient Recruiting — https://www.bmsstudyconnect.com/s/US/English/USenHome
- See also: Investigator Inquiry Form — https://www.bms.com/researchers-and-partners/investigator-inquiry-form.html
- See also: FDA Safety Alerts and Recalls — https://www.fda.gov/Safety/MedWatch/SafetyInformation/default.htm

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 10 participants randomized and treated
Groups:
- Arm A (Part 1): BMS-986277 IV 3 X 10^10
  Cycle 1 of BMS-986277 will be administered as a single IV infusion (D1) before proceeding to sequential dosing (consisting of 3 doses administered on Days 15, 17, and 19). A minimum of 24 hours is required between doses of BMS-986277.
- Arm B (Part 1): BMS-986277 IV 3 X 10^11
  Cycle 1 of BMS-986277 will be administered as a single IV infusion (D1) before proceeding to sequential dosing (consisting of 3 doses administered on Days 15, 17, and 19). A minimum of 24 hours is required between doses of BMS-986277.
- Arm C (Part 1): BMS-986277 IV 1 X 10^12
  Cycle 1 of BMS-986277 will be administered as a single IV infusion (D1) before proceeding to sequential dosing (consisting of 3 doses administered on Days 15, 17, and 19). A minimum of 24 hours is required between doses of BMS-986277.
Period: Overall Study
Arm/Group | Arm A (Part 1) | Arm B (Part 1) | Arm C (Part 1)
Started (Started = Entering the treatment period) | 4 | 3 | 3
Completed (Completed = Completing the treatment period) | 1 | 0 | 1
Not Completed | 3 | 3 | 2
Not completed — Progressive disease | 2 | 3 | 1
Not completed — Study drug toxicity | 0 | 0 | 1
Not completed — Death | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Arm A (Part 1) | Arm B (Part 1) | Arm C (Part 1) | Total
Number analyzed (Participants) | 4 | 3 | 3 | 10
Age, Continuous [Mean (Standard Deviation); unit: Years] | 61 (2.4) | 59 (10.4) | 47 (12.1) | 57 (9.9)
Age, Customized [Count of Participants; unit: Participants]
  > 65 years | 0 | 1 | 0 | 1
  <= 65 years | 4 | 2 | 3 | 9
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 1 | 2 | 5
  Male | 2 | 2 | 1 | 5
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0 | 0
  Not Hispanic or Latino | 1 | 0 | 1 | 2
  Unknown or Not Reported | 3 | 3 | 2 | 8
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0
  White | 4 | 3 | 3 | 10
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With an Adverse Event (AE)
Description: Number of participants who experienced an AE during the course of the study.
Time Frame: from first dose to 60 days post last dose, assessed up to February 2020 (approx. 26 months)
Population: All treated participants
  Study terminated, data not reported due to privacy reasons
Measure: Number; unit: Number of Participants
Arm/Group | Arm A (Part 1) | Arm B (Part 1) | Arm C (Part 1)
Number analyzed (Participants) | 4 | 3 | 3
Number of Participants | NA — Study terminated, data not reported due to privacy reasons | NA — Study terminated, data not reported due to privacy reasons | NA — Study terminated, data not reported due to privacy reasons

2. Primary Outcome: Number of Participants With a Serious Adverse Event (SAE)
Description: Number of participants who experienced a SAE during the course of the study.
Time Frame: from first dose to 60 days post last dose, assessed up to February 2020 (approx. 26 months)
Population: All treated participants
  Study terminated, data not reported due to privacy reasons
Measure: Number; unit: Number of Participants
Arm/Group | Arm A (Part 1) | Arm B (Part 1) | Arm C (Part 1)
Number analyzed (Participants) | 4 | 3 | 3
Number of Participants | NA — Study terminated, data not reported due to privacy reasons | NA — Study terminated, data not reported due to privacy reasons | NA — Study terminated, data not reported due to privacy reasons

3. Primary Outcome: Number of Participants With an Adverse Event (AE) Meeting Protocol-defined Dose Limiting Toxicity (DLT) Criteria
Description: Number of participants who experienced an AE meeting protocol-defined DLT criteria during the course of the study.
Time Frame: from first dose to 60 days post last dose, assessed up to February 2020 (approx. 26 months)
Population: All treated participants
  Study terminated, data not reported due to privacy reasons
Measure: Number; unit: Number of Participants
Arm/Group | Arm A (Part 1) | Arm B (Part 1) | Arm C (Part 1)
Number analyzed (Participants) | 4 | 3 | 3
Number of Participants | NA — Study terminated, data not reported due to privacy reasons | NA — Study terminated, data not reported due to privacy reasons | NA — Study terminated, data not reported due to privacy reasons

4. Primary Outcome: Number of Participants With an Adverse Event (AE) Leading to Discontinuation
Description: Number of participants who experienced an AE leading to discontinuation during the course of the study.
Time Frame: from first dose to 60 days post last dose, assessed up to February 2020 (approx. 26 months)
Population: All treated participants
  Study terminated, data not reported due to privacy reasons
Measure: Number; unit: Number of Participants
Arm/Group | Arm A (Part 1) | Arm B (Part 1) | Arm C (Part 1)
Number analyzed (Participants) | 4 | 3 | 3
Number of Participants | NA — Study terminated, data not reported due to privacy reasons | NA — Study terminated, data not reported due to privacy reasons | NA — Study terminated, data not reported due to privacy reasons

5. Primary Outcome: Number of Participants With an Adverse Event (AE) Leading to Death
Description: Number of participants who experienced an AE leading to death during the course of the study.
Time Frame: from first dose to 60 days post last dose, assessed up to February 2020 (approx. 26 months)
Population: All treated participants
  Study terminated, data not reported due to privacy reasons
Measure: Number; unit: Number of Participants
Arm/Group | Arm A (Part 1) | Arm B (Part 1) | Arm C (Part 1)
Number analyzed (Participants) | 4 | 3 | 3
Number of Participants | NA — Study terminated, data not reported due to privacy reasons | NA — Study terminated, data not reported due to privacy reasons | NA — Study terminated, data not reported due to privacy reasons

6. Primary Outcome: Number of Participants With a Clinical Laboratory Test Abnormality
Description: Number of participants who experienced a clinical laboratory test abnormality during the course of the study.
Time Frame: from first dose to 60 days post last dose, assessed up to February 2020 (approx. 26 months)
Population: All treated participants
  Study terminated, data not reported due to privacy reasons
Measure: Number; unit: Number of Participants
Arm/Group | Arm A (Part 1) | Arm B (Part 1) | Arm C (Part 1)
Number analyzed (Participants) | 4 | 3 | 3
Number of Participants | NA — Study terminated, data not reported due to privacy reasons | NA — Study terminated, data not reported due to privacy reasons | NA — Study terminated, data not reported due to privacy reasons

7. Primary Outcome: Number of Participants With a Vital Sign Abnormality or Other Safety Biomarkers
Description: Number of participants who experienced a vital sign abnormality or other safety biomarkers during the course of the study.
Time Frame: from first dose to 60 days post last dose, assessed up to February 2020 (approx. 26 months)
Population: All treated participants
  Study terminated, data not reported due to privacy reasons
Measure: Number; unit: Number of Participants
Arm/Group | Arm A (Part 1) | Arm B (Part 1) | Arm C (Part 1)
Number analyzed (Participants) | 4 | 3 | 3
Number of Participants | NA — Study terminated, data not reported due to privacy reasons | NA — Study terminated, data not reported due to privacy reasons | NA — Study terminated, data not reported due to privacy reasons

8. Secondary Outcome: Objective Response Rate (ORR)
Description: ORR is defined as the proportion of all treated participants whose BOR is either CR or PR. BOR was determined by investigators for the reported data.
  Estimate of ORR and corresponding 2-sided exact 95% CI using the Clopper-Pearson method
Time Frame: at Weeks 8, 16 and 24
Population: All treated participants
  Study terminated, data not reported due to privacy reasons
Measure: Number; unit: Percentage of Participants
Arm/Group | Arm A (Part 1) | Arm B (Part 1) | Arm C (Part 1)
Number analyzed (Participants) | 4 | 3 | 3
Percentage of Participants | NA — Study terminated, data not reported due to privacy reasons | NA — Study terminated, data not reported due to privacy reasons | NA — Study terminated, data not reported due to privacy reasons

9. Secondary Outcome: Disease Control Rate (DCR)
Description: DCR includes complete response (CR), partial response (PR), and stable disease (SD).
  Estimate of DCR and corresponding 2-sided exact 95% CI using the Clopper-Pearson method
Time Frame: at Weeks 8, 16 and 24
Population: All treated participants
  Study terminated, data not reported due to privacy reasons
Measure: Number; unit: Percentage of Participants
Arm/Group | Arm A (Part 1) | Arm B (Part 1) | Arm C (Part 1)
Number analyzed (Participants) | 4 | 3 | 3
Percentage of Participants | NA — Study terminated, data not reported due to privacy reasons | NA — Study terminated, data not reported due to privacy reasons | NA — Study terminated, data not reported due to privacy reasons

10. Secondary Outcome: Median Duration of Response (mDOR)
Description: DOR for a participant with a BOR of CR or PR is defined as the time between the date of first response and the date of the first objectively documented tumor progression per RECIST v1.1/PCWG3 or death, whichever occurs first.
  Estimate by the Kaplan-Meier method and corresponding 2-sided 95% CI using Brookmeyer and Crowley methodology (using log-log transformation)
Time Frame: at Weeks 8, 16 and 24
Population: All treated participants
  Study terminated, data not reported due to privacy reasons
Measure: Number; unit: Number of Participants
Arm/Group | Arm A (Part 1) | Arm B (Part 1) | Arm C (Part 1)
Number analyzed (Participants) | 4 | 3 | 3
Number of Participants | NA — Study terminated, data not reported due to privacy reasons | NA — Study terminated, data not reported due to privacy reasons | NA — Study terminated, data not reported due to privacy reasons

11. Secondary Outcome: Median Progression-Free Survival (mPFS)
Description: PFS for a participant is defined as the time from the first dosing date to the date of first objectively documented disease progression or death due to any cause, whichever occurs first.
  Estimate by the Kaplan-Meier method and corresponding 2-sided 95% CI using Brookmeyer and Crowley methodology (using log-log transformation) for the median and Greenwood formula for the rate.
Time Frame: at Weeks 8, 16 and 24, to progression
Population: All treated participants
  Study terminated, data not reported due to privacy reasons
Measure: Number; unit: Number of Participants
Arm/Group | Arm A (Part 1) | Arm B (Part 1) | Arm C (Part 1)
Number analyzed (Participants) | 4 | 3 | 3
Number of Participants | NA — Study terminated, data not reported due to privacy reasons | NA — Study terminated, data not reported due to privacy reasons | NA — Study terminated, data not reported due to privacy reasons

12. Secondary Outcome: Progression-Free Survival Rate (PFSR)
Description: as for outcome 11
Time Frame: at Weeks 8, 16 and 24
Population: All treated participants
  Study terminated, data not reported due to privacy reasons
Measure: Number; unit: Percentage of Participants
Arm/Group | Arm A (Part 1) | Arm B (Part 1) | Arm C (Part 1)
Number analyzed (Participants) | 4 | 3 | 3
Percentage of Participants | NA — Study terminated, data not reported due to privacy reasons | NA — Study terminated, data not reported due to privacy reasons | NA — Study terminated, data not reported due to privacy reasons

13. Secondary Outcome: Cmax
Description: Pharmacokinetics of BMS-986277 were derived from blood concentration versus time data.
  Cmax is defined as the maximum observed blood concentration.
Time Frame: Cycle 1 (Day 1 pre-dose through Day 29, 240 hour), Cycle 2 (Day 1 pre-dose through Day 22, 408 hour); through Follow-up visits
Population: All treated participants
  Study terminated, data not reported due to privacy reasons
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: µg/mL
Arm/Group | Arm A (Part 1) | Arm B (Part 1) | Arm C (Part 1)
Number analyzed (Participants) | 4 | 3 | 3
µg/mL | NA (NA) — Study terminated, data not reported due to privacy reasons | NA (NA) — Study terminated, data not reported due to privacy reasons | NA (NA) — Study terminated, data not reported due to privacy reasons

14. Secondary Outcome: Tmax
Description: Pharmacokinetics of BMS-986277 were derived from blood concentration versus time data.
  Tmax is defined as the time of maximum observed blood concentration.
Time Frame: as for outcome 13
Population: All treated participants
  Study terminated, data not reported due to privacy reasons
Measure: Median (Full Range); unit: hour
Arm/Group | Arm A (Part 1) | Arm B (Part 1) | Arm C (Part 1)
Number analyzed (Participants) | 4 | 3 | 3
hour | NA [NA to NA] — Study terminated, data not reported due to privacy reasons | NA [NA to NA] — Study terminated, data not reported due to privacy reasons | NA [NA to NA] — Study terminated, data not reported due to privacy reasons

15. Secondary Outcome: AUC(0-T)
Description: Pharmacokinetics of BMS-986277 were derived from blood concentration versus time data.
  AUC(0-T) is the area under the blood concentration-time curve from time zero to time of last quantifiable concentration.
Time Frame: as for outcome 13
Population: All treated participants
  Study terminated, data not reported due to privacy reasons
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: µg.h/mL
Arm/Group | Arm A (Part 1) | Arm B (Part 1) | Arm C (Part 1)
Number analyzed (Participants) | 4 | 3 | 3
µg.h/mL | NA (NA) — Study terminated, data not reported due to privacy reasons | NA (NA) — Study terminated, data not reported due to privacy reasons | NA (NA) — Study terminated, data not reported due to privacy reasons

16. Secondary Outcome: AUC(INF)
Description: Pharmacokinetics of BMS-986277 were derived from blood concentration versus time data.
  AUC(INF) is the area under the blood concentration-time curve from time zero extrapolated to infinite time.
Time Frame: as for outcome 13
Population: All treated participants
  Study terminated, data not reported due to privacy reasons
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: µg.h/mL
Arm/Group | Arm A (Part 1) | Arm B (Part 1) | Arm C (Part 1)
Number analyzed (Participants) | 4 | 3 | 3
µg.h/mL | NA (NA) — Study terminated, data not reported due to privacy reasons | NA (NA) — Study terminated, data not reported due to privacy reasons | NA (NA) — Study terminated, data not reported due to privacy reasons

17. Secondary Outcome: T-HALF
Description: Pharmacokinetics of BMS-986277 were derived from blood concentration versus time data.
  T-HALF is defined as the apparent terminal half-life.
Time Frame: as for outcome 13
Population: All treated participants
  Study terminated, data not reported due to privacy reasons
Measure: Mean (Standard Deviation); unit: hour
Arm/Group | Arm A (Part 1) | Arm B (Part 1) | Arm C (Part 1)
Number analyzed (Participants) | 4 | 3 | 3
hour | NA (NA) — Study terminated, data not reported due to privacy reasons | NA (NA) — Study terminated, data not reported due to privacy reasons | NA (NA) — Study terminated, data not reported due to privacy reasons

18. Secondary Outcome: CLT
Description: Pharmacokinetics of BMS-986277 were derived from blood concentration versus time data.
  CLT is defined as the total body clearance.
Time Frame: as for outcome 13
Population: All treated participants
  Study terminated, data not reported due to privacy reasons
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: liter
Arm/Group | Arm A (Part 1) | Arm B (Part 1) | Arm C (Part 1)
Number analyzed (Participants) | 4 | 3 | 3
liter | NA (NA) — Study terminated, data not reported due to privacy reasons | NA (NA) — Study terminated, data not reported due to privacy reasons | NA (NA) — Study terminated, data not reported due to privacy reasons

19. Secondary Outcome: Vss
Description: Pharmacokinetics of BMS-986277 were derived from blood concentration versus time data.
  Vss is defined as the volume of distribution at steady-state.
Time Frame: as for outcome 13
Population: All treated participants
  Study terminated, data not reported due to privacy reasons
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: liter
Arm/Group | Arm A (Part 1) | Arm B (Part 1) | Arm C (Part 1)
Number analyzed (Participants) | 4 | 3 | 3
liter | NA (NA) — Study terminated, data not reported due to privacy reasons | NA (NA) — Study terminated, data not reported due to privacy reasons | NA (NA) — Study terminated, data not reported due to privacy reasons

20. Secondary Outcome: Vz
Description: Pharmacokinetics of BMS-986277 were derived from blood concentration versus time data.
  Vz is defined as the volume of distribution of the elimination phase.
Time Frame: as for outcome 13
Population: All treated participants
  Study terminated, data not reported due to privacy reasons
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: liter
Arm/Group | Arm A (Part 1) | Arm B (Part 1) | Arm C (Part 1)
Number analyzed (Participants) | 4 | 3 | 3
liter | NA (NA) — Study terminated, data not reported due to privacy reasons | NA (NA) — Study terminated, data not reported due to privacy reasons | NA (NA) — Study terminated, data not reported due to privacy reasons

21. Secondary Outcome: AUC(0-48)
Description: Pharmacokinetics of BMS-986277 were derived from blood concentration versus time data.
  AUC(0-T) is the area under the blood concentration-time curve from time zero to 48 hours postdose
Time Frame: Cycle 1 (from time zero to 48 hours postdose)
Population: All treated participants
  Study terminated, data not reported due to privacy reasons
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: µg.h/mL
Arm/Group | Arm A (Part 1) | Arm B (Part 1) | Arm C (Part 1)
Number analyzed (Participants) | 4 | 3 | 3
µg.h/mL | NA (NA) — Study terminated, data not reported due to privacy reasons | NA (NA) — Study terminated, data not reported due to privacy reasons | NA (NA) — Study terminated, data not reported due to privacy reasons

22. Secondary Outcome: AUC(0-8)
Description: Pharmacokinetics of BMS-986277 were derived from blood concentration versus time data.
  AUC(0-T) is the area under the blood concentration-time curve from time zero to 8 hours postdose
Time Frame: Cycle 1 (from time zero to 8 hours postdose)
Population: All treated participants
  Study terminated, data not reported due to privacy reasons
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: µg.h/mL
Arm/Group | Arm A (Part 1) | Arm B (Part 1) | Arm C (Part 1)
Number analyzed (Participants) | 4 | 3 | 3
µg.h/mL | NA (NA) — Study terminated, data not reported due to privacy reasons | NA (NA) — Study terminated, data not reported due to privacy reasons | NA (NA) — Study terminated, data not reported due to privacy reasons

23. Secondary Outcome: C48
Description: Pharmacokinetics of BMS-986277 were derived from blood concentration versus time data.
  C48 is defined as the blood concentration at 48 hours postdose.
Time Frame: Cycle 1 at 48 hours postdose
Population: All treated participants
  Study terminated, data not reported due to privacy reasons
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: µg/mL
Arm/Group | Arm A (Part 1) | Arm B (Part 1) | Arm C (Part 1)
Number analyzed (Participants) | 4 | 3 | 3
µg/mL | NA (NA) — Study terminated, data not reported due to privacy reasons | NA (NA) — Study terminated, data not reported due to privacy reasons | NA (NA) — Study terminated, data not reported due to privacy reasons

24. Secondary Outcome: Css-avg
Description: Pharmacokinetics of BMS-986277 were derived from blood concentration versus time data.
  Css-avg is defined as the average blood concentration over a dosing interval at steady state (AUC[0-48]/48).
Time Frame: Cycle 1 (from time zero to 48 hours postdose)
Population: All treated participants
  Study terminated, data not reported due to privacy reasons
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: µg/mL
Arm/Group | Arm A (Part 1) | Arm B (Part 1) | Arm C (Part 1)
Number analyzed (Participants) | 4 | 3 | 3
µg/mL | NA (NA) — Study terminated, data not reported due to privacy reasons | NA (NA) — Study terminated, data not reported due to privacy reasons | NA (NA) — Study terminated, data not reported due to privacy reasons

25. Secondary Outcome: AI_AUC
Description: Pharmacokinetics of BMS-986277 were derived from blood concentration versus time data.
  AUC accumulation index; ratio of AUC(0-48) on Cycle 1 Day 19 to AUC(0-48) on Cycle 1 Day 15 for monotherapy.
Time Frame: Cycle 1 (Day 19, Day 15)
Population: All treated participants
  Study terminated, data not reported due to privacy reasons
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ratio AUC(0-48),C1D19 to AUC(0-48),C1D15
Arm/Group | Arm A (Part 1) | Arm B (Part 1) | Arm C (Part 1)
Number analyzed (Participants) | 4 | 3 | 3
ratio AUC(0-48),C1D19 to AUC(0-48),C1D15 | NA (NA) — Study terminated, data not reported due to privacy reasons | NA (NA) — Study terminated, data not reported due to privacy reasons | NA (NA) — Study terminated, data not reported due to privacy reasons

26. Secondary Outcome: AI_Cmax
Description: Pharmacokinetics of BMS-986277 were derived from blood concentration versus time data.
  Cmax accumulation index; ratio of Cmax on Cycle 1 Day 19 to Cmax on Cycle 1 Day 15 for monotherapy.
Time Frame: Cycle 1 (Day 19, Day 15)
Population: All treated participants
  Study terminated, data not reported due to privacy reasons
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ratio of Cmax,C1D19 to Cmax,C1D15
Arm/Group | Arm A (Part 1) | Arm B (Part 1) | Arm C (Part 1)
Number analyzed (Participants) | 4 | 3 | 3
ratio of Cmax,C1D19 to Cmax,C1D15 | NA (NA) — Study terminated, data not reported due to privacy reasons | NA (NA) — Study terminated, data not reported due to privacy reasons | NA (NA) — Study terminated, data not reported due to privacy reasons

27. Secondary Outcome: T-HALFeff
Description: Pharmacokinetics of BMS-986277 were derived from blood concentration versus time data.
  T-HALFeff is defined as effective elimination half-life that explains the degree of accumulation observed for a specific exposure measure (exposure measure includes AUC, Cmax)
Time Frame: as for outcome 13
Population: All treated participants
  Study terminated, data not reported due to privacy reasons
Measure: Median (Full Range); unit: hour
Arm/Group | Arm A (Part 1) | Arm B (Part 1) | Arm C (Part 1)
Number analyzed (Participants) | 4 | 3 | 3
hour | NA [NA to NA] — Study terminated, data not reported due to privacy reasons | NA [NA to NA] — Study terminated, data not reported due to privacy reasons | NA [NA to NA] — Study terminated, data not reported due to privacy reasons

28. Secondary Outcome: Ctrough
Description: Pharmacokinetics of BMS-986277 were derived from blood concentration versus time data.
  Ctrough is defined as the trough observed blood concentration.
Time Frame: as for outcome 13
Population: All treated participants
  Study terminated, data not reported due to privacy reasons
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: µg/mL
Arm/Group | Arm A (Part 1) | Arm B (Part 1) | Arm C (Part 1)
Number analyzed (Participants) | 4 | 3 | 3
µg/mL | NA (NA) — Study terminated, data not reported due to privacy reasons | NA (NA) — Study terminated, data not reported due to privacy reasons | NA (NA) — Study terminated, data not reported due to privacy reasons

29. Secondary Outcome: Number of Participants With a Positive Antibody-Drug-Antibody (ADA) Response
Description: Baseline ADA-positive participant is defined as a participant who has an ADA-detected sample at baseline.
  ADA-positive participant is a participant with at least 1 ADA-positive sample relative to baseline after initiation of the treatment.
  Frequency distribution of baseline ADA-positive participants and ADA-positive participants after initiation of the treatment
Time Frame: as for outcome 13
Population: All treated participants
  Study terminated, data not reported due to privacy reasons
Measure: Number; unit: Number of participants
Arm/Group | Arm A (Part 1) | Arm B (Part 1) | Arm C (Part 1)
Number analyzed (Participants) | 4 | 3 | 3
Number of participants | NA — Study terminated, data not reported due to privacy reasons | NA — Study terminated, data not reported due to privacy reasons | NA — Study terminated, data not reported due to privacy reasons

ADVERSE EVENTS:
Time Frame: AEs/SAEs are collected from the first dose date until the last dose date + 100 days, assessed up to February 2020 (approx. 26 months)
Arm/Group | Arm A (Part 1) | Arm B (Part 1) | Arm C (Part 1)
All-Cause Mortality (participants affected / at risk) | 2/4 | 2/3 | 2/3
Serious Adverse Events (participants affected / at risk) | 1/4 | 0/3 | 2/3
Other Adverse Events (participants affected / at risk) | 4/4 | 3/3 | 3/3
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Arm A (Part 1) (N=4) | Arm B (Part 1) (N=3) | Arm C (Part 1) (N=3)
Ascites (Gastrointestinal disorders) | 1 | 0 | 0
Cytokine release syndrome (Immune system disorders) | 0 | 0 | 1
Dehydration (Metabolism and nutrition disorders) | 0 | 0 | 1
Malignant neoplasm progression (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 2
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Arm A (Part 1) (N=4) | Arm B (Part 1) (N=3) | Arm C (Part 1) (N=3)
Abdominal distension (Gastrointestinal disorders) | 1 | 0 | 0
Abdominal pain (Gastrointestinal disorders) | 1 | 1 | 0
Abdominal pain lower (Gastrointestinal disorders) | 0 | 1 | 0
Constipation (Gastrointestinal disorders) | 1 | 0 | 0
Diarrhoea (Gastrointestinal disorders) | 2 | 0 | 0
Dry mouth (Gastrointestinal disorders) | 0 | 0 | 1
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 1 | 1 | 0
Haemorrhoidal haemorrhage (Gastrointestinal disorders) | 1 | 0 | 0
Lip ulceration (Gastrointestinal disorders) | 1 | 0 | 0
Nausea (Gastrointestinal disorders) | 3 | 1 | 2
Stomatitis (Gastrointestinal disorders) | 0 | 0 | 1
Vomiting (Gastrointestinal disorders) | 1 | 1 | 2
Chills (General disorders) | 1 | 1 | 2
Fatigue (General disorders) | 2 | 1 | 3
Influenza like illness (General disorders) | 0 | 2 | 0
Oedema peripheral (General disorders) | 0 | 0 | 1
Pyrexia (General disorders) | 0 | 0 | 3
Cytokine release syndrome (Immune system disorders) | 0 | 1 | 1
Urinary tract infection (Infections and infestations) | 1 | 0 | 0
Alanine aminotransferase increased (Investigations) | 1 | 0 | 0
Amylase increased (Investigations) | 0 | 1 | 0
Aspartate aminotransferase increased (Investigations) | 1 | 1 | 0
Blood bilirubin increased (Investigations) | 1 | 0 | 0
Blood creatinine increased (Investigations) | 0 | 1 | 0
Lipase increased (Investigations) | 0 | 1 | 0
Decreased appetite (Metabolism and nutrition disorders) | 2 | 1 | 0
Hypomagnesaemia (Metabolism and nutrition disorders) | 0 | 1 | 0
Hypophosphataemia (Metabolism and nutrition disorders) | 0 | 1 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 1 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 2
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 1 | 1
Neck pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Headache (Nervous system disorders) | 1 | 2 | 1
Sciatica (Nervous system disorders) | 0 | 1 | 0
Insomnia (Psychiatric disorders) | 1 | 0 | 0
Hypertonic bladder (Renal and urinary disorders) | 1 | 0 | 0
Micturition urgency (Renal and urinary disorders) | 1 | 0 | 0
Haematospermia (Reproductive system and breast disorders) | 0 | 1 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Productive cough (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Hot flush (Vascular disorders) | 0 | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less

DOCUMENTS (2):
  • Study Protocol (2018-08-15): https://cdn.clinicaltrials.gov/large-docs/76/NCT03363776/Prot_000.pdf
  • Statistical Analysis Plan (2018-03-12): https://cdn.clinicaltrials.gov/large-docs/76/NCT03363776/SAP_001.pdf